CLINICAL TRIAL: NCT06599437
Title: Index Laparoscopic Cholecystectomy Following Clearance of Common Bile Duct Stones Via Endoscopic Retrograde Cholangiography
Brief Title: For Patients with Stones in Gallbladder and Bile Duct Stones At the Same Time, Surgical Removal of the Gallbladder with the Laparoscope is Done in the Same Admission Compared to Its Removal After 6 Weeks Following Successful Removel of the Stones from the Bile Ducts by the Side View Endoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour Medical National Institute (Other Government)
Responsible Party: Principal Investigator, Wael Ahmed El-Dawy, Lecturer of Hepatopacreatobiliary and GI Surgery, Damanhour Medical National Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HD000192
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Choledocholithiasis with Cholecystitis
Keywords: choledocholithiasis; ERCP; Early cholecystectomy
MeSH Terms: conditions — Choledocholithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early same admission laparoscopic cholecystectomy ( group A) (Active Comparator): Early laparoscopic cholecystectomy is performed on next day within 24 hours after common bile duct stone removal by ERCP.
  Interventions: Procedure: laparoscopic cholecystectomy
- Late laparoscopic cholecystectomy ( group B) (Active Comparator): Late laparoscopic cholecystectomy is performed 6 weeks after common bile duct stones clearance
  Interventions: Procedure: Late laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy — Early laparoscopic cholecystectomy in the same admission after atone clearance from the bile ducts via ERCP.
  Arms: Early same admission laparoscopic cholecystectomy ( group A)
Procedure: Late laparoscopic cholecystectomy — Laparoscopic cholecystectomy is performed 6 weeks after clearance of stones from the common bile duct.
  Arms: Late laparoscopic cholecystectomy ( group B)

SUMMARY:
The goal of this clinical trial is to learn if early laparoscopic cholecystectomy is safe and feasible when performed during the same admission for patients with concomitant gallbladder and common bile duct stones after clearance of CBD stones via ERCP in comparison to Late laparoscopic cholecystectomy 6 weeks after ERCP. The main questions it aims to answer are: laparoscopic cholecystectomy

* Does index laparoscopic cholecystectomy associate with less recurrence of biliary complications?
* Is index laparoscopic cholecystectomy feasible and safe for the patients in terms of intraoperative difficulties, conversion to open, hospital stay, and postoperative complications than late laparoscopic cholecystectomy? the investigator will compare index laparoscopic cholecystectomy with late laparoscopic cholecystectomy 6 weeks after ERCP to see if index laparoscopic cholecystectomy is safe and feasible and associated with better outcomes.

Participants will:

Come to the outpatient clinic every week after intervention for follow-up for 3 months after surgery.

DETAILED DESCRIPTION:
The study population of this randomized controlled trial study is those who underwent CBD stone clearance by ERCP. The included fifty patients were stratified randomly into two groups: early and delayed.

Randomization was done using computer-generated random number sequences in concealed envelopes with a block randomization design. Laparoscopic cholecystectomy is performed on the next day after successful clearance of stones from CBD while, the patient is still admitted, for the early group and postponed 4 to 6 weeks for the delayed group after the patient is discharged home.

Laparoscopic cholecystectomy was performed by the same surgical team for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with concomitant gallbladder and common bile duct stone who underwent clearance of common bile duct stones by ERCP

Exclusion Criteria: patients with any of the following:

* Severe pancreatitis
* Suspicion of post-ERCP bleeding or perforation,
* Associated malignancy
* Those in whom ERCP failed to clear the CBD stones

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
recurrence of biliary events | up to 3 months after surgery
  the occurence of acute cholecystitism biliary colics, common bile duct stonem pancreatitisand cholangitis after ERCP while waiting for laparoscopic cholecystectomy

SECONDARY OUTCOMES:
operative time | during surgery
  time from the first incision of skin to skin closure and completion of surgery
pancreatitis | 3 months after surgery
  acute inflammation of the pancreas : abdominal pain, elevated lipase and amylase ( more than 3 folds) and/or findings specific for the pancreatitits on imaging.
conversion to open surgery | During surgery
  termination of the laparoscopic procedure and perfome the surgery by the conventional open surgery
Bleeding | during surger and up to 3 weeks
  Intraoperative or postoperative bleeding that requires blood transfusion
the presence of intraoperative adhesions | During surgery
  Adhesions around the gallbladder and at the Calot's triangle
Bile leak | up to 1 week after surgery
  the leak of bile through the drain or intraabdominally
Wound infection | up to 3 months after surgery
  Any evidence of infection in the wounds : redness, pain or discharge of infected fluids from the wounds
hospital stays | from admission to the end of post operative follow up at 3 months after surgery
  the sum the length of stay after ERCP and laparoscopic cholecystectomy including readmission for complication management
post oprative pain | after surgery and up to 3 days
  the degree pain described by the patients after surgery on the visual rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Damanhur Medical National Institute, Damanhur, Behira, Egypt